CLINICAL TRIAL: NCT03724643
Title: Protocolized Ventilator Weaning Verses Usual Care: A Randomized Controlled Trial
Brief Title: Protocolized Ventilator Weaning Verses Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, PhD, Senior Intensivist Nurse, Baqiyatallah Medical Sciences University, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BUMS-PWvUC-RCT
Record Dates: First submitted 2018-10-04; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Failure
Keywords: Mechanical ventilation; Ventilator weaning; Extubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protocolized Wean (Experimental): Respiratory therapist determined extubation readiness based on: patent and protected airway; adequate secretion clearance; suction requirement ≤ every 2 hours; FiO2 < 50% and PEEP = 5; and hemodynamic stability without circulatory support. The SBT included CPAP = 5 mmHg at FiO2 ≤ 0.4. Patients were assessed after 3-minutes for appropriateness to continue (SaO2 ≥ 92%; no arrhythmia; RSBI < 105 breaths/min/L). Respiratory distress signs included RR > 30 breaths/min, SaO2< 90%, HR > 140 beats/min, or a sustained change in HR of >20%, systolic BP >200 mmHg or <80 mmHg, or agitation, anxiety, or diaphoresis without other cause. The SBT lasted 120 min in accordance with prior studies. Upon SBT completion, the RSBI was re-measured and an ABG was obtained.
  Interventions: Other: Protocolized wean
- Usual Care (No Intervention): In the UC group, the SBT type and extubation decision was determined by the attending intensivist on service based upon neurologic status, airway competence (gag, cough, suction requirements), and negative inspiratory force (NIF) or RSBI measurements.

INTERVENTIONS:
Other: Protocolized wean — Respiratory therapist determined extubation readiness based on: patent and protected airway; adequate secretion clearance; suction requirement ≤ every 2 hours; FiO2 < 50% and PEEP = 5; and hemodynamic stability without circulatory support. The SBT included CPAP = 5 mmHg at FiO2 ≤ 0.4. Patients were assessed after 3-minutes for appropriateness to continue (SaO2 ≥ 92%; no arrhythmia; RSBI < 105 breaths/min/L). Respiratory distress signs included RR > 30 breaths/min, SaO2< 90%, HR > 140 beats/min, or a sustained change in HR of >20%, systolic BP >200 mmHg or <80 mmHg, or agitation, anxiety, or diaphoresis without other cause. The SBT lasted 120 min in accordance with prior studies. Upon SBT completion, the RSBI was re-measured and an ABG was obtained.
  Arms: Protocolized Wean

SUMMARY:
Protocol-driven ventilator weaning strategies utilizing spontaneous breathing trials (SBT) reportedly result in shorter intubation duration and intensive care unit (ICU) length-of-stay (LOS). Investigators compared respiratory therapy (RT)-driven protocolized ventilator weaning (PW) verses usual care (UC) as it pertains to physiologic respiratory parameters, intubation duration, extubation success/reintubation rates, and ICU LOS. The study was a prospective multicenter randomized controlled trial in 6 ICUs at 6 academic-affiliated hospitals in a resource limited setting. Extubation readiness was determined by the attending physician (UC) or the respiratory therapist (PW) using pre-defined criteria and SBT. Physiologic variables, serial blood gas measurements, and weaning indices were assessed including rapid shallow breathing index (RSBI), negative inspiratory force (NIF), occlusion pressure (P0.1), dynamic and static compliance (Cdyn and Cs).

DETAILED DESCRIPTION:
This was a prospective multicenter randomized controlled trial in 6 closed ICUs with 24/7 in-house intensivist coverage at 6 academic-affiliated medical centers in a resource limited setting from October 18, 2007 to May 03, 2014. All parts of the study were reviewed according to the Consolidated Standards for Reporting Trials (CONSORT) statement. Crossover was not allowed. Participants were blinded to randomization group, as were the healthcare providers and statistician. Randomization was accomplished using Random Allocation Software© (RAS; Informer Technologies, Inc.). Block randomization was performed by a computer generated random number list prepared by a statistician. Allocation consignment occurred through confidential communication between the patient's nurse and a third party not involved in recruitment. The data analyzer was blinded to group randomization and was not present during ventilator weaning. There were no important changes to methods after trial commencement. The study ended because it achieved the necessary sample size.

Pparticipants were randomly assigned to ventilator weaning either by protocolized methodology or by usual care (UC). All patients were ventilated using Dräger Evita® XL or Evita® 4 ventilators (Dräeger Medical, Inc., Lubeck, Germany). In the PW group, weaning and extubation readiness was determined by the RT using pre-defined criteria and the result of a SBT. Pre-defined weaning criteria included: (1) patent upper airway; (2) ability to protect airway (defined by mental status and presence of adequate gag and cough reflexes); (3) ability to clear secretions; (4) decreasing secretion burden requiring suction not more frequently than every 2 hours; (5) level of support (FiO2 < 50%, PEEP = 5); and (6) hemodynamic stability not requiring chemical (vasopressors, inotropes) or mechanical (e.g. intra-aortic balloon pump, extracorporeal life support) circulatory support. Until the SBT, management of each group was the same. For patients in the UC group, SBT type and determination to extubate was determined by attending physician preference. For participants in the PW group, the SBT type was protocol determined, and extubation decisions were driven by RT. The SBT consisted of continuous positive airway pressure (CPAP) of 5 mmHg with an FiO2 ≤ 0.4. After 3-minutes patients were assessed for appropriateness to continue the SBT by arterial oxygen saturation (SaO2) ≥ 92% without arrhythmias, and a rapid shallow breathing index (RSBI = RR/VT) < 105 breaths/min/L. Specified signs of respiratory distress included respiratory rate (RR)> 30 breaths/minute, SaO2< 90%, heart rate (HR)> 140 breaths/minute, or a sustained increase or decrease of HR of >20%, systolic blood pressure >200 mmHg or <80 mmHg, or agitation, anxiety, or diaphoresis without other identified cause. The SBT was performed for 120 min in accordance with prior studies. At the end of the SBT, the RSBI was re-measured and an arterial blood gas (ABG) was obtained.

In the UC group, the SBT type and extubation decision was determined by the attending intensivist on service based upon neurologic status, airway competence (gag, cough, suction requirements), and negative inspiratory force (NIF) or RSBI measurements. Extubation success was defined as remaining extubated for 48 hours without need for re-intubation or other forms of non-invasive MV.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ICU
* Endotracheally intubated on mechanical ventilation ≥ 24 hours
* Full-code status
* Informed consent provided by the patient, legal guardian, or healthcare surrogate (prior to ventilator weaning).

Exclusion Criteria:

* Declining consent
* Death without ventilator weaning
* Cardiopulmonary arrest on the ventilator
* Permanent ventilator dependence
* Tracheostomy placement for long-term weaning
* Self-extubation
* Pulmonary edema
* Aspiration during the wean
* Copious secretions and mucus plugging precluding wean
* Severe obstructive lung disease
* COPD with hypercapneic respiratory failure
* Status-post-respiratory arrest
* Concurrent neurologic / neuromuscular comorbidity
* Drug or alcohol intoxication
* Incomplete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4200 (Actual)
Dates: Start 2007-10-18 (Actual); Primary Completion 2014-05-03 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
Duration of Intubation | through study completion, an average of 30 days
  Duration of mechanical ventilation

SECONDARY OUTCOMES:
Hospital length-of-stay | through study completion, an average of 30 days
  Hospital length-of-stay

IPD SHARING:
Plan to Share IPD: Undecided